CLINICAL TRIAL: NCT05041439
Title: Adherence to Care for Children Born to Mothers With Laboratory Evidence of Confirmed or Possible Congenital Zika Virus Infection During Pregnancy.
Brief Title: Adherence to Care for Children With Congenital Zika Virus Infection in Puerto Rico
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Puerto Rico (Other)
Responsible Party: Principal Investigator, Julie H Levison, Assistant Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021p001675; 5R21HD096369-02 (NIH)
Record Dates: First submitted 2021-09-02; First posted 2021-09-13 (Actual); Results first posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-11

CONDITIONS: Zika Virus Infection; Adherence, Patient
Keywords: Zika virus; Puerto Rico; community health worker
MeSH Terms: conditions — Zika Virus Infection; Patient Compliance | interventions — Community Health Workers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community health worker (CHW) group (Experimental): Participants in the intervention arm will receive 5 one-on-one sessions over 6 months with a CHW, as well as a manual and written materials on child development. At baseline and exit, all participants will be assessed using instruments to measure demographics and self-perceived barriers.
  Interventions: Behavioral: Community Health Worker
- Enhanced care condition (ECC) (No Intervention): Participants in this arm will receive 5 outreach calls at the same interval as the intervention arm, as well as written materials on child development. At baseline and exit, all participants will be assessed using instruments to measure demographics and self-perceived barriers.

INTERVENTIONS:
Behavioral: Community Health Worker — Participants will receive 5 one-on-one sessions with a CHW over 6 months.
  Arms: Community health worker (CHW) group

SUMMARY:
Given the magnitude of the epidemic in Puerto Rico, congenital Zika virus infection may have devastating complications to a significant population of children, also affecting families and society at large. This proposal takes a critical first step to ensuring that children with exposure to congenital Zika virus infection receive the follow-up care they need for optimal clinical outcomes. We anticipate that lessons learned from this study may also positively impact models for adherence to early intervention services in Puerto Rico.

DETAILED DESCRIPTION:
Overview:

Participants will be the primary caregivers (age ≥18 years) of children with possible congenital Zika virus infection. Participants will be recruited from the pediatric services of the University of Puerto Rico Medical Sciences Campus (UPR-MSC), as well as other clinics and community-based organizations in Puerto Rico. In the intervention, a community health worker (CHW) will deliver personalized sessions framed around a multi-media health communication tool. The CHW will deliver the intervention over a 6-month period.

Study procedures:

Participants will be the primary caregivers (age ≥18 years) of children with possible congenital Zika virus infection. Participants will be recruited via provider referral, peer referral, and flyers. Once an individual expresses interest in the study, a study staff member will screen that individual to assess eligibility. Individuals who are eligible will be invited to enroll through an informed consent process and complete a baseline interview. After completion of the baseline interview, study staff will randomize participants into an enhanced control condition (ECC) or intervention condition that receives an individually-tailored community health worker intervention. At trial exit, all participants, including the ECC group, will complete an in-depth assessment to measure their barriers to follow-up Zika-related pediatric services and provide feedback about their experience in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older and able to communicate in Spanish
* Being the primary caregiver of a child with possible congenital Zika virus infection

Exclusion Criteria:

* Those who are too sick/unable to understand the implications of their participation, those who are unwilling to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie H. Levison, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- School of Medicine - Department of Pediatrics, San Juan, PR, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 60 participants were screened for eligibility and 50 were consented/enrolled.
Period: Overall Study
Arm/Group | Community Health Worker (CHW) Group | Enhanced Care Condition (ECC)
Started | 25 | 25
Completed | 23 | 24
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Community Health Worker (CHW) Group | Enhanced Care Condition (ECC) | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (7.6) | 30.2 (5.9) | 32.6 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 25 | 50
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Amerian Indian | 1 | 0 | 1
  Black | 1 | 4 | 5
  White | 4 | 0 | 4
  Multiracial | 12 | 13 | 25
  Other | 6 | 7 | 13
  Unknown | 1 | 1 | 2
Baseline sociodemographic and clinical characteristics of randomized participants [Count of Participants; unit: Participants] | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adherence to Pediatric Zika Care
Description: At least one pediatric visit for developmental exam with the pediatrician within 6 months post-randomization.
Time Frame: Within the first 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Community Health Worker (CHW) Group | Enhanced Care Condition (ECC)
Number analyzed (Participants) | 25 | 25
Participants | 14 | 15

2. Secondary Outcome: Number of Participants With Detection of Zika-associated Birth Defect or Neurodevelopmental Abnormality
Description: Detection of new birth defect or neurodevelopmental abnormality between baseline to month-6.
Time Frame: Within the first 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Community Health Worker (CHW) Group | Enhanced Care Condition (ECC)
Number analyzed (Participants) | 25 | 25
Participants | 1 | 3

3. Secondary Outcome: Number of Participants With Adherence to Pediatric Zika Care
Description: At least two pediatric visits recorded within 12 months post-randomization, with one visit from months 0-6 and months 7-12.
Time Frame: Within the first 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Community Health Worker (CHW) Group | Enhanced Care Condition (ECC)
Number analyzed (Participants) | 25 | 25
Participants | 6 | 5

4. Secondary Outcome: Number of Participants With Detection of Zika-associated Birth Defect or Neurodevelopmental Abnormality
Description: Detection of new birth defect or neurodevelopmental abnormality between baseline to month-12.
Time Frame: Within the first 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Community Health Worker (CHW) Group | Enhanced Care Condition (ECC)
Number analyzed (Participants) | 25 | 25
Participants | 1 | 4

ADVERSE EVENTS:
Time Frame: The monitoring for adverse events was over the 12 months of the study.
Arm/Group | Community Health Worker (CHW) Group | Enhanced Care Condition (ECC)
All-Cause Mortality (participants affected / at risk) | 1/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Community Health Worker (CHW) Group (N=25) | Enhanced Care Condition (ECC) (N=25)
Complications of diabetes (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/39/NCT05041439/Prot_SAP_000.pdf